CLINICAL TRIAL: NCT06977451
Title: An Open-Label Single Center, Single Participant Study of an Experimental Antisense Oligonucleotide Treatment for Amyotrophic Lateral Sclerosis (ALS) Due to an Arg15Leu Pathogenic Variant in CHCHD10
Brief Title: Personalized Antisense Oligonucleotide for a Single Participant With CHCHD10 ALS
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: n-Lorem Foundation (Other)
Collaborators: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAV1774
Record Dates: First submitted 2025-05-09; First posted 2025-05-18 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-05

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open Label (Experimental)
  Interventions: Drug: nL-CHCHD-001

INTERVENTIONS:
Drug: nL-CHCHD-001 — Personalized Antisense Oligonucleotide

SUMMARY:
This research project entails delivery of a personalized antisense oligonucleotide (ASO) drug designed for a single participant with amyotrophic lateral sclerosis (ALS) due to a pathogenic variant in CHCHD10

ELIGIBILITY:
Inclusion Criteria:

* Informed consent/assent provided by the participant (when appropriate), and/or participant's parent(s) or legally authorized representative(s).
* Ability to travel to the study stie and adhere to study-related follow-up examinations and/or procedures and provide access to participant's medical records.
* Genetically confirmed neurological disorder.

Exclusion Criteria:

* Participant has any condition that in the opinion of the Site Investigator, would ultimately prevent the completion of study procedures.
* Use of an investigational medication within less than 5 half-lives of the drug at enrollment

Ages: 63 Years to 63 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2024-06-24 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Clinical Functioning | Baseline to 12 months
  Change from baseline at 12-months post nL-CHCHD-001 administration in scores on Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised (ALSFRS-R). A maximum score of 48 represents normal functioning, and the minimum score is 0.
Motor Functioning | Baseline to 12 months
  Change from baseline at 12-months post nL-CHCHD-001 administration in scores on Slow Vital Capacity (SVC) Performance.
Motor Functioning | Baseline to 12 months
  Change from baseline at 12-months post nL-CHCHD-001 administration in scores on Handheld Dynamometry (HHD).
Clinical Functioning | Baseline to 12 months
  Change from baseline at 12-months post nL-CHCHD-001 administration in scores on Edinburgh Cognitive and Behavioral ALS Screen (ECAS).
Clinical Functioning | Baseline to 12 months
  Change from baseline at 12-months post nL-CHCHD-001 administration in scores on ALS Cognitive Behavioral Screen (ALS-CBS)
Clinical Functioning | Baseline to 12 months
  Change from baseline at 12-months post nL-CHCHD-001 administration in scores on Amyotrophic Lateral Sclerosis Assessment Questionnaire 5 (ALSAQ-5)

SECONDARY OUTCOMES:
Disease Biomarkers | Baseline to 12 months
  Change from baseline at 12-months post nL-CHCHD-001 administration in serum and cerebrospinal fluid neurofilament light chain levels
Safety and Tolerability | Baseline to 12 months
  Incidence and Severity of Adverse Events
Safety and Tolerability | Baseline to 12 months
  Emergent abnormalities in physical exam
Safety and Efficacy | Baseline to 12 months
  Emergent abnormalities in neurological exam
Safety and Efficacy | Baseline to 12 months
  Emergent abnormalities in safety labs (CSF, chemistry, hematology, coagulation, and urinalysis)

CONTACTS AND LOCATIONS:
Locations (1):
- Columbia University, Irving Medical Center, New York, New York, United States